CLINICAL TRIAL: NCT00637312
Title: Clinical Trial Comparing the Blackstone Advent™ Cervical Disc to Anterior Cervical Discectomy and Fusion (ACDF) for the Treatment of One Level Degenerative Disc Disease
Brief Title: Advent™ Cervical Disc Versus ACDF for Treatment of One Level Degenerative Disc Disease (IDE Study)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Greater-than-anticipated rate of revisions
Sponsor: Orthofix Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CP-01003
Record Dates: First submitted 2008-03-10; First posted 2008-03-17 (Estimated); Results first posted 2014-03-27 (Estimated); Last update posted 2014-03-27 (Estimated); Status verified 2014-02

CONDITIONS: Cervical Degenerative Disc Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Advent™ Cervical Disc (Experimental): Cervical artificial disc replacement: Advent™ Cervical Disc
  Interventions: Device: Cervical Artificial Disc (Advent™ Cervical Disc)
- Standard care - Control (Active Comparator): Anterior cervical discectomy and fusion (ACDF) with Hallmark™ Anterior Cervical Plate System
  Interventions: Device: Hallmark™ Anterior Cervical Plate System

INTERVENTIONS:
Device: Cervical Artificial Disc (Advent™ Cervical Disc) — Advent™ Cervical Disc
  Other Names: Advent™ Cervical Disc
  Arms: Advent™ Cervical Disc
Device: Hallmark™ Anterior Cervical Plate System — Hallmark™ Anterior Cervical Plate System with AlloQuent Structural Allograft (corticocancellous allograft bone)
  Arms: Standard care - Control

SUMMARY:
The purpose of this study is to establish the safety and effectiveness of the Advent™ Cervical Disc compared to Anterior Cervical Discectomy and Fusion (ACDF) in treating degenerative disc disease at a single-level in the cervical spine (from C3 to C7) following cervical discectomy in skeletally mature patients (at least 18 years of age).

DETAILED DESCRIPTION:
Following surgery study subjects will be evaluated at the following intervals: 6 wks (± 2wks); 3 Months (±2 wks); 6 Month (±1 months); 12 and 24 Month (±2 months) and annually until the last subject enrolled completes their 24 Month follow-up

ELIGIBILITY:
Inclusion Criteria:

* One cervical spine level between C3 and C7 which requires surgical treatment for intractable cervical radiculopathy and/or myelopathy demonstrated by herniated disc, and/or osteophyte formation leading to nerve root and/or spinal cord compression confirmed by patient history (e.g. neck and/or arm pain), functional and/or neurological deficit (e.g. numbness, weakness, diminished or pathologic reflexes, gait disturbances, etc.) and radiographic studies (e.g. CT, MRI, x-rays, etc.).
* Unresponsive to conservative care over a period of at least 6 weeks
* Neck Disability Index score ≥ 15/50 (30%)
* Willing and able to comply with the requirements of the protocol including follow-up requirements and to sign a study specific informed consent

Exclusion Criteria:

* More than 1 level requiring surgical treatment for intractable cervical radiculopathy and/or myelopathy.
* Active local (at the proposed surgical site) or systemic infection
* Prior anterior neck surgery at any level.
* Prior posterior cervical spine surgery at the index level except posterior decompressive surgery where the posterior elements are preserved.
* Currently undergoing treatment for disease of the thoracic or lumbar spine.
* Axial neck pain as the primary diagnosis, without evidence of neural compression
* Significant cervical anatomical deformity
* Any anatomical consideration which in the investigators opinion would make the anterior cervical approach excessively risky or impossible
* Severe obesity defined as a Body Mass Index (BMI) > 40
* Instability on AP, lateral neutral or flex/ext images: ≥2mm translation relative to the adjacent segment, and/or ≥ 11 degrees relative to adjacent segments
* Central disc height ≤ 2mm
* Advanced spondylosis (i.e. facet joints degeneration, anterior or posterior bridging of the interspace or lack of motion on the pre-operative flexion/extension x-rays)
* Severe cervical myelopathy as indicated by: Signs and/or symptoms > 6months duration, Nurick's Classification grades IV or V, and/or Myelomalacia as evidence on a MRI
* Metabolic bone disease such as osteoporosis to a degree that spinal instrumentation is contra-indicated (Males over 55 years of age, females over 50 years of age and/or subjects that in the investigators opinion are medical indicative of osteoporosis (e.g. early menopause, steroid use, etc.) are required to have a DEXA scan; If the DEXA scan is ≤ -2.5t in the spine, the patient must be excluded)
* Allergy to any component of the device (titanium, polycarbonated polyurethane, polyethylene terephthalate, or ethylene oxide residuals)
* Chronic steroid or other medication use that may interfere with bony/soft tissue healing
* History of endocrine or metabolic disorders (e.g. Paget's disease) known to effect bone and mineral metabolism
* Autoimmune diseases e.g., ankylosing spondylitis, rheumatoid arthritis, etc.
* Insulin dependent diabetes mellitus
* Active malignancy
* Currently pregnant or considering becoming pregnant during the follow-up period
* Advanced emphysema, Alzheimer's disease or other medical conditions that would interfere with patient self-assessment of function, pain or quality of life
* Medical condition (e.g. unstable cardiac disease, end-stage cancer) that may result in patient death prior to study completion
* Chemical dependency (e.g. alcohol or narcotic addiction) problem that may interfere with study requirements
* Mental incompetence as determined by the Investigator which may effect participation in the study
* Incarcerated
* Involved in any current or pending litigation relating to a spinal condition
* Concurrently participating in any other investigational study
* Anatomy (e.g. endplate dimensions) at the index level not consistent with the dimensions of the implants available (e.g. based on pre-operative radiographic evaluations and templates in the surgical technique manual).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2008-03; Primary Completion 2011-07 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott L Blumenthal, M.D., Study Director — Texas Back Institute
Locations (13):
- United States (13):
  - University of California Davis, Sacramento, California
  - Boulder Neurosurgical Associates, Boulder, Colorado
  - University of South Florida, Tampa, Florida
  - Spine Institute of Louisiana, Shreveport, Louisiana
  - Brain and Spine Specialist, Baltimore, Maryland
  - Cooper University Neurological Institute, Camden, New Jersey
  - University of Rochester Medical Center, Rochester, New York
  - Triangle Orthopaedics Associates, P.A., Durham, North Carolina
  - University of Pennsylvania, Department of Neurosurgery, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - East Tennessee Brain and Spine Center, Johnson City, Tennessee
  - Texas Back Institute, Plano, Texas
  - The San Antonio Orthopaedic Group, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Advent™ Cervical Disc | Standard Care - Control
Started | 72 | 36
Completed | 30 | 19
Not Completed | 42 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Advent™ Cervical Disc | Standard Care - Control | Total
Number analyzed (Participants) | 72 | 36 | 108
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 72 | 36 | 108
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43 (8.5) | 45.6 (9.1) | 43.9 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 19 | 55
  Male | 36 | 17 | 53
Region of Enrollment [Number; unit: participants]
  United States | 72 | 36 | 108

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of Device and/or Procedure Related Adverse Event(s)
Time Frame: At 24-months
Population: The study was suspended for higher than anticipated adverse events in the treatment group. Enrollment was stopped and patients were followed for 36 months in the Advent treatment group. Agency approval is not being pursued for this device and thus no analysis has been completed.
Arm/Group | Advent™ Cervical Disc | Standard Care - Control
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected immediately post-op through the 24 month visit for control patients and through 36 months for treatment patients.
Description: Adverse events were collected at all routine and unscheduled follow-up visits.
Arm/Group | Advent™ Cervical Disc | Standard Care - Control
Serious Adverse Events (participants affected / at risk) | 16/72 | 1/36
Other Adverse Events (participants affected / at risk) | 58/72 | 21/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Advent™ Cervical Disc (N=72) | Standard Care - Control (N=36)
Medical device removal (Surgical and medical procedures) | 16 (17) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Advent™ Cervical Disc (N=72) | Standard Care - Control (N=36)
Neck Pain (Musculoskeletal and connective tissue disorders) | 26 (26) | 8 (8)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 20 (20) | 10 (10)
Pseudoarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
Back Pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 5 (5)
Exostosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Muscle strain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 12 (12) | 4 (4)
Paraesthesia (Nervous system disorders) | 5 (5) | 4 (4)
Headache (Nervous system disorders) | 9 (9) | 4 (4)
Burning sensation (Nervous system disorders) | 2 (2) | 0 (0)
Muscular weakness (Nervous system disorders) | 2 (2) | 1 (1)
Nervous system disorder (Nervous system disorders) | 2 (2) | 0 (0)
Dysaesthesia (Nervous system disorders) | 0 (0) | 2 (2)
Hemiparesis (Nervous system disorders) | 0 (0) | 1 (1)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Intervertebral disc operation (Surgical and medical procedures) | 1 (1) | 1 (1)
Pain (General disorders) | 3 (3) | 1 (1)
Herpes zoster (Infections and infestations) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 0 (0)
Anxiety postoperative (Psychiatric disorders) | 0 (0) | 1 (1)
Procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Urinary retention postoperative (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Eyelid ptosis (Eye disorders) | 0 (0) | 1 (1)
Hypothyroidism (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was suspended for a high rate of adverse events in the treatment group. Enrollment was stopped and patients were followed for 36 months in the Advent group. Approval is not being pursued and thus no analysis has been completed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Within the first 12 months following completion of the study, any publication must be initiated as a multi-center publication in conjunction with other PIs in the study. After 12 months, each PI is able to publish their data, but must first submit the publication to the sponsor within 60 days prior to publication. The sponsor has the right to make reasonable requests to protect the rights and interests of the sponsor.